CLINICAL TRIAL: NCT02055157
Title: A Phase 2, Open-label, Sequential Cohort Dose-escalation Study of BMN 111 in Children With Achondroplasia
Brief Title: A Phase 2 Study of BMN 111 to Evaluate Safety, Tolerability, and Efficacy in Children With Achondroplasia
Acronym: ACH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 111-202; 2013-004137-32 (EudraCT Number)
Record Dates: First submitted 2013-04-18; First posted 2014-02-05 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism; Bone Diseases, Developmental; Bone Diseases
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases, Developmental; Bone Diseases | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Cohort 1: 2.5 ug/kg
  Interventions: Drug: BMN 111
- Cohort 2 (Experimental): Cohort 2: 7.5 ug/kg,
  Interventions: Drug: BMN 111
- Cohort 3 (Experimental): Cohort 3: 15 ug/Kg
  Interventions: Drug: BMN 111
- Cohort 4 (Experimental): Cohort 4: 30 ug/kg
  Interventions: Drug: BMN 111

INTERVENTIONS:
Drug: BMN 111 — BMN 111 will be administered daily for 24 months in an open-label sequential dose adjustment fashion.
  Other Names: Modified recombinant human C-type natriuretic peptide; Vosoritide

SUMMARY:
This is a Phase 2, open-label, sequential cohort dose-escalation study of BMN 111 in children with achondroplasia. The primary objective is to assess the safety and tolerability of daily BMN 111 administered to children with achondroplasia.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or guardian(s) are willing and able to provide written, signed informed consent
* 5 to 14 years old at end of study
* ACH, documented by clinical grounds, confirmed by genetic testing
* At least 6-month of pretreatment growth assessment in Study 111-901 before study entry, and one standing height at least 6 months prior to screening for 111-202
* Negative pregnancy test at the Screening Visit for females ≥ 10 years old or who have begun menses
* If sexually active, willing to use a highly effective method of contraception while participating in the study
* Ambulatory, able to stand without assistance
* Willing and able to perform all study procedures as physically possible
* Parents/caregivers willing to administer daily injections to the subjects

Additional inclusion Criteria Optional, Open-label Extension Phase:

* Appropriate written informed consent

Exclusion Criteria:

* Hypochondroplasia or short stature condition other than ACH
* Have any of the following:

  * Hypothyroidism or hyperthyroidism
  * Insulin-requiring diabetes mellitus
  * Autoimmune inflammatory disease
  * Inflammatory bowel disease
  * Autonomic neuropathy
  * Recent acute illness associated with volume dehydration not completely resolved prior to the first dose of study drug
* Unstable condition requiring surgical intervention during the study
* Growth plates have fused
* Have a history of any of the following:

  * Renal insufficiency, defined as creatinine > 2 mg/dl
  * Anemia
  * Baseline systolic BP < 75 mm Hg or recurrent symptomatic hypotension or recurrent symptomatic hypotension, recurrent symptomatic orthostatic hypotension
  * Cardiac or vascular disease, including the following:

    * Cardiac dysfunction (abnormal echocardiogram [ECHO] including left ventricle [LV] mass) at Screening Visit
    * Hypertrophic cardiomyopathy
    * Pulmonary Hypertension
    * Congenital heart disease with ongoing cardiac dysfunction
    * Cerebrovascular disease
    * Aortic insufficiency
    * Clinically significant atrial or ventricular arrhythmias
* Have an ECG showing any of the following:

  * Right or left atrial enlargement or ventricular hypertrophy
  * PR (period of time from the beginning of atrial depolarization until the beginning of ventricular depolarization) interval > 200 msec
  * QRS (The Q, R, and S heart waves that are measured on an electrocardiogram) interval > 110 msec
  * Corrected QTc-F (Measure of the corrected time between the start of the Q wave and end of the T wave in the heart's electrical cycle) > 450 msec
  * Second- or third-degree atrioventricular block
* Documented Vitamin D deficiency
* Require any investigational agent prior to completion of study period
* Have received another investigational product or investigational medical device within 30 days before the Screening visit
* Use of any other investigational product or investigational medical device for the treatment of ACH or short stature
* Current chronic therapy with antihypertensive medications, angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, diuretics, beta-blockers, calcium-channel blockers, cardiac glycosides, systemic anticholinergic agents, any medication that may impair or enhance compensatory tachycardia, diuretics, or other drugs known to alter renal or tubular function
* Treatment with growth hormone, IGF-1 (Insulin-like growth factor), or anabolic steroids in the previous 6 months or long-term treatment (> 3 months) at any time
* Long-term treatment (> 1 month) with oral corticosteroids
* Concomitant medication that prolongs the QT/QTc-F interval within 14 days or 5 half-lives, whichever is longer, before the Screening visit
* Pregnant or breastfeeding at the Screening Visit or planning to become pregnant (self or partner) at any time during the study
* Limb-lengthening or bone-related surgery < 18 months prior to study enrollment
* Had a fracture of the long bones or spine within 6 months prior to screening (except for fracture of digits or toes)
* AST (Aspartate Transaminase) or ALT (Alanine Transaminase) at least 3x upper limit of normal (ULN) or total bilirubin at least 2x ULN
* Evidence of severe sleep apnea requiring surgery or new initiation of CPAP (Continuous positive airway pressure).
* History of malignancy and chemotherapy/radiation or currently under work-up for suspected malignancy
* Known hypersensitivity to BMN 111 or its excipients
* Have a condition or circumstance that, in the view of the Investigator, places the subject at high risk for poor treatment compliance or for not completing the study
* Concurrent disease or condition that would interfere with study participation or safety
* Have abnormal findings on baseline clinical hip exam or imaging assessments that are determined to be clinically significant as determined by the PI.
* Have a history of hip surgery or severe hip dysplasia
* Have a history of clinically significant hip injury in the 30 days prior to screening.
* History of slipped capital femoral epiphysis or avascular necrosis of the femoral head.
* Are unable to lie flat when in prone position

Additional Exclusion Criteria for Optional, Open-label Extension Phase:

* Use of restricted therapies during the initial 6 months of the study
* Permanently discontinued BMN 111 during the initial 6 months of the study

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (9):
- United States (6):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins McKusick - Institute of Genetic Medicine, Baltimore, Maryland
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Institut Necker, Paris, France
- Guys & St. Thomas NHS Foundation Trust Evelina Hospital, London, United Kingdom

REFERENCES:
- [Derived] Qi Y, Chan ML, Mould DR, Larimore K, Fisheleva E, Cherukuri A, Day J, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Bober MB, Henshaw J. Development of a Weight-Band Dosing Approach for Vosoritide in Children with Achondroplasia Using a Population Pharmacokinetic Model. Clin Pharmacokinet. 2024 May;63(5):707-719. doi: 10.1007/s40262-024-01371-6. Epub 2024 Apr 23. PMID 38649657
- [Derived] Chan ML, Qi Y, Larimore K, Cherukuri A, Seid L, Jayaram K, Jeha G, Fisheleva E, Day J, Huntsman-Labed A, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Horton WA, Henshaw J. Pharmacokinetics and Exposure-Response of Vosoritide in Children with Achondroplasia. Clin Pharmacokinet. 2022 Feb;61(2):263-280. doi: 10.1007/s40262-021-01059-1. Epub 2021 Aug 25. PMID 34431071
- [Derived] Savarirayan R, Irving M, Bacino CA, Bostwick B, Charrow J, Cormier-Daire V, Le Quan Sang KH, Dickson P, Harmatz P, Phillips J, Owen N, Cherukuri A, Jayaram K, Jeha GS, Larimore K, Chan ML, Huntsman Labed A, Day J, Hoover-Fong J. C-Type Natriuretic Peptide Analogue Therapy in Children with Achondroplasia. N Engl J Med. 2019 Jul 4;381(1):25-35. doi: 10.1056/NEJMoa1813446. Epub 2019 Jun 18. PMID 31269546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at nine study centers in United States, Australia, United Kingdom and France.
Groups:
- Cohort 1: Initial 6 months: BMN 111 at 2.5 μg/kg daily subcutaneous injection, over a period of 6 months.
  18-month extension: BMN 111 at 2.5 μg/kg daily subcutaneous injection, dose determined to be suboptimal after the end of the initial 6 months, 7 subjects escalated to 7.5 μg/kg daily subcutaneous injection, discontinued 1 subject escalating 6 subjects to BMN 111 at 15.0 μg/kg daily subcutaneous injection, over a period of 18 months.
- Cohort 2: Initial 6 months: BMN 111 at 7.5 μg/kg daily subcutaneous injection, over a period of 6 months.
  18-month extension: BMN 111 at 7.5 μg/kg daily subcutaneous injection, dose determined to be suboptimal after the end of the initial 6 months, discontinued 1 subject escalating 6 subjects to BMN 111 at 15.0 μg/kg daily subcutaneous injection, over a period of 18 months.
- Cohort 3: Initial 6 months: BMN 111 at 15.0 μg/kg daily subcutaneous injection, over a period of 6 months.
  18-month extension: BMN 111 at 15.0 μg/kg daily subcutaneous injection, over a period of 18 months.
- Cohort 4: Initial 6 months: BMN 111 at 30.0 μg/kg daily subcutaneous injection, over a period of 6 months.
  18-month extension: BMN 111 at 30.0 μg/kg daily subcutaneous injection, over a period of 18 months.
Period: Initial 6 Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 8 | 8 | 10 | 9
Completed | 7 | 7 | 10 | 8
Not Completed | 1 | 1 | 0 | 1
Not completed — Subject discontinued due to NeedlePhobia | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Consent withdrawn by subject | 1 | 0 | 0 | 0
Period: 18-month Extension
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 7 | 7 | 10 | 8
Completed | 6 | 6 | 10 | 8
Not Completed | 1 | 1 | 0 | 0
Not completed — Investigator decision | 0 | 1 | 0 | 0
Not completed — Subject discontinued due to NeedlePhobia | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population consists of all subjects who received at least one dose of study treatment and were used for safety analysis in the initial 6-month period and entire study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 8 | 8 | 10 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: yrs] | 7.3 (1.58) | 8.3 (2.19) | 8.0 (1.63) | 6.9 (1.17) | 7.6 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 5 | 19
  Male | 3 | 5 | 4 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 8 | 9 | 7 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 6 | 5 | 6 | 24
  Asian | 0 | 1 | 3 | 3 | 7
  Black or African American | 1 | 0 | 1 | 0 | 2
  Other | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Adverse Events During Initial 6-Month Period
Description: A treatment-emergent Adverse Events (TEAE) is any Adverse Events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration.
  Serious adverse event (SAE).
Time Frame: Up to Month 6 ± 7 Days
Population: Safety Analysis Population includes all subjects who received at least one dose of study treatment and were used for safety analysis in the initial 6-month period and entire study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 9
Participants
  Subjects with at Least 1 Reported TEAE | 8 | 8 | 10 | 9
  Subjects Least Reported Study Drug-Related TEAE | 7 | 8 | 9 | 9
  Subjects with at Least 1 Reported SAE | 0 | 0 | 0 | 0
  Subjects Least Reported Study Drug-Related SAE | 0 | 0 | 0 | 0
  Subjects Who Died | 0 | 0 | 0 | 0

2. Primary Outcome: Overall Summary of Adverse Events During Entire Study Period
Description: A treatment-emergent Adverse Events (TEAE) is any Adverse Events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration.
  TEAE - Treatment-emergent adverse event. SAE - Serious adverse event.
Time Frame: Up to Month 25 ± 7 Days
Population: Safety Analysis Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 9
Participants
  Subjects with at Least 1 Reported TEAE | 8 | 8 | 10 | 9
  Subjects Least Reported Study Drug-Related TEAE | 7 | 8 | 9 | 9
  Subjects with at Least 1 Reported SAE | 1 | 0 | 1 | 1
  Subjects Least Reported Study Drug-Related SAE | 0 | 0 | 0 | 0
  Subjects Who Died | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Annualized Growth Velocity (AGV) During Initial 6-Month
Description: Annualized Growth Velocity at Day 183 is assessed on standing height as ((Height at Day 183 Visit - Height at Baseline Visit)/(Date at Day 183 Visit - Baseline Visit Date)) x 365.25.
Time Frame: At 6 month (Day 183)
Population: Efficacy Analysis Population includes all subjects who received at least one dose of study treatment and who had post treatment data for any efficacy endpoint in the corresponding period were included in the Efficacy Analysis and Extension Efficacy Analysis population.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
cm/year
  Baseline | 3.755 (1.1094) | 2.891 (1.3920) | 4.044 (2.2751) | 4.492 (1.1889)
  Change from Baseline to Day 183: number analyzed (Participants) | 7 | 8 | 10 | 8
  Change from Baseline to Day 183 | -0.371 (1.5920) | 1.276 (1.4387) | 2.014 (1.9990) | 2.085 (2.1375)

4. Secondary Outcome: Change From Baseline in Annualized Growth Velocity (AGV) During Entire Study Period - Cohort 3 and 4
Description: Annualized Growth Velocity at Day 183 visit is assessed on standing height as ((Height at Day 183 Visit - Height at Baseline Visit)/(Date at Day 183 Visit - Baseline Visit Date)) x 365.25.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
cm/year
  Baseline | 4.044 (2.2751) | 4.492 (1.1889)
  Change from Baseline to Month 24 | 1.744 (1.7974) | 1.538 (1.3387)

5. Secondary Outcome: Change From Baseline in Annualized Growth Velocity (AGV) During Entire Study Period - Cohort 1 and 2 Switchers
Description: Annualized Growth Velocity at 1st visit with >= 12 months on 15ug/kg is assessed on standing height as ((Height at 1st Visit with >= 12 Months on 15 μg/kg - Height at 1st Visit on 15 μg/kg)/(Date of the 1st Visit with >= 12 months on 15 μg/kg - Date of at 1st Visit on 15 μg/kg)) x 365.25.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
cm/year
  Baseline | 3.629 (1.1586) | 3.510 (0.8327)
  Change from Baseline at >=12 Months on 15μg/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline at >=12 Months on 15μg/kg | 1.846 (2.1466) | 2.245 (0.9176)

6. Secondary Outcome: Change From Baseline in Height Z-Scores Using Centers for Disease Control and Prevention (CDC) Reference Standard During Initial 6-Months
Description: Height Z scores indicates how far a particular child is from the average height for children of the same sex and age. A positive height Z score indicates the child's height is above average whilst a negative Z score indicates the child's height is below average. Height Z scores below -2 Standard Deviation Scores (SDs) indicate a child's height is no longer within normal height range for average stature children of the same sex and age.
  Z-scores are derived using non-ACH age-sex-specific reference data (means and standard deviations) per Centers for Disease Control and Prevention (CDC).
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
z score
  Baseline: number analyzed (Participants) | 7 | 8 | 10 | 8
  Baseline | -6.056 (0.6331) | -5.145 (0.8530) | -4.613 (1.1355) | -5.193 (0.7486)
  Change from Baseline to Day 183: number analyzed (Participants) | 7 | 8 | 10 | 8
  Change from Baseline to Day 183 | -0.008 (0.1788) | 0.078 (0.1440) | 0.229 (0.1505) | 0.265 (0.1869)

7. Secondary Outcome: Change From Baseline in Height Z-Scores Using CDC Reference Standard During Entire Study Period - Cohort 3 and 4
Description: Height Z scores indicates how far a particular child is from the average height for children of the same sex and age. A positive height Z score indicates the child's height is above average whilst a negative Z score indicates the child's height is below average. Height Z scores below -2 SDs indicate a child's height is no longer within normal height range for average stature children of the same sex and age.
  Z-scores are derived using non-ACH age-sex-specific reference data (means and standard deviations) per Centers for Disease Control and Prevention (CDC).
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
z score
  Baseline | -4.613 (1.1355) | -5.193 (0.7486)
  Change from Baseline to Month 24 | 0.788 (0.2842) | 0.896 (0.3010)

8. Secondary Outcome: Change From Baseline in Height Z-Scores Using CDC Reference Standard During Entire Study Period - Cohort 1 and 2 Switchers
Description: as for outcome 7
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
z score
  Baseline | -6.064 (0.6932) | -4.912 (0.7708)
  Change from Baseline to >=12 Months on 15ug/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline to >=12 Months on 15ug/kg | 0.520 (0.2950) | 0.259 (0.1887)

9. Secondary Outcome: Change From Baseline in Upper to Lower Body Ratios During Initial 6-Months
Description: The Upper to Lower Body ratio prior to treatment, at baseline, and through 6 months is assessed on Sitting Height / (Standing Height - Sitting Height)
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
Ratio
  Baseline: number analyzed (Participants) | 7 | 8 | 10 | 8
  Baseline | 2.094 (0.0984) | 2.027 (0.1793) | 1.911 (0.2286) | 1.962 (0.1822)
  Change from Baseline to Day 183: number analyzed (Participants) | 7 | 8 | 10 | 8
  Change from Baseline to Day 183 | -0.021 (0.0626) | 0.003 (0.0510) | -0.024 (0.0369) | -0.030 (0.0811)

10. Secondary Outcome: Change From Baseline in Upper to Lower Body Ratios During Entire Study Period - Cohort 3 and 4
Description: The Upper to Lower Body ratio prior to treatment, at baseline, and through 24 months is assessed on Sitting Height / (Standing Height - Sitting Height)
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
ratio
  Baseline | 1.911 (0.2286) | 1.962 (0.1822)
  Change from Baseline to Month 24 | -0.067 (0.0451) | -0.121 (0.1058)

11. Secondary Outcome: Change From Baseline in Upper Arm Length to Lower Arm (Forearm) Length Ratio During Initial 6-Months
Description: The Upper Arm Length to Lower Arm (Forearm) Length ratio prior to treatment, at baseline, and through 6 months is assessed on Upper Arm Length / Lower Arm (Forearm) Length.
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
ratio
  Baseline: number analyzed (Participants) | 7 | 8 | 10 | 8
  Baseline | 1.130 (0.1168) | 1.143 (0.0924) | 1.130 (0.1190) | 1.106 (0.0816)
  Change from Baseline to Day 183 | -0.019 (0.0623) | 0.001 (0.0521) | -0.048 (0.1002) | 0.003 (0.0869)

12. Secondary Outcome: Change From Baseline in Upper Arm to Lower Arm Length Ratio During Entire Study Period - Cohort 3 and 4
Description: The Upper Arm Length to Lower Arm (Forearm) Length ratio prior to treatment, at baseline, and through 24 months is assessed on Upper Arm Length / Lower Arm (Forearm) Length.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
ratio
  Baseline | 1.130 (0.1190) | 1.106 (0.0816)
  Change from Baseline to Month 24 | 0.037 (0.0673) | -0.027 (0.0504)

13. Secondary Outcome: Change From Baseline in Upper to Lower Body Ratios During Entire Study Period - Cohort 1 and 2 Switchers
Description: as for outcome 10
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
ratio
  Baseline | 2.119 (0.0812) | 2.053 (0.1746)
  Change from Baseline to >=12 Months on 15ug/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline to >=12 Months on 15ug/kg | -0.078 (0.0452) | -0.078 (0.1271)

14. Secondary Outcome: Change From Baseline in Upper Arm to Lower Arm Length Ratio During Entire Study Period - Cohort 1 and 2 Switchers
Description: as for outcome 12
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
ratio
  Baseline | 1.131 (0.1280) | 1.114 (0.0520)
  Change from Baseline to >=12 Months on 15ug/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline to >=12 Months on 15ug/kg | 0.009 (0.0056) | -0.004 (0.1181)

15. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Knee to Heel Length Ratio During Initial 6-months
Description: The Upper Leg Length (Thigh) to Knee to Heel Length Ratio prior to treatment, at baseline, and through 6 months is assessed on Upper Leg Length (Thigh) / Knee to Heel Length.
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
ratio
  Baseline: number analyzed (Participants) | 7 | 8 | 10 | 8
  Baseline | 0.672 (0.0600) | 0.662 (0.0585) | 0.687 (0.0268) | 0.691 (0.0847)
  Change from Baseline to Day 183: number analyzed (Participants) | 7 | 8 | 10 | 8
  Change from Baseline to Day 183 | -0.002 (0.0401) | -0.006 (0.0462) | 0.007 (0.0411) | -0.006 (0.0810)

16. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Knee to Heel Length Ratio During Entire Study Period - Cohort 3 and 4
Description: The Upper Leg Length (Thigh) to Knee to Heel Length Ratio prior to treatment, at baseline, and through 24 months is assessed by Upper Leg Length (Thigh) / Knee to Heel Length.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
ratio
  Baseline | 0.687 (0.0268) | 0.691 (0.0847)
  Change from Baseline to Month 24 | 0.010 (0.0503) | -0.033 (0.1065)

17. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Knee to Heel Length Ratio During Entire Study Period - Cohort 1 and 2 Switchers
Description: as for outcome 16
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
ratio
  Baseline | 0.659 (0.0541) | 0.673 (0.0579)
  Change from Baseline to >=12 Months on 15ug/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline to >=12 Months on 15ug/kg | 0.002 (0.0228) | 0.006 (0.0618)

18. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Tibial Length Ratio During Initial 6-months
Description: The Upper Leg Length (Thigh) to Tibial Length Ratio prior to treatment, at baseline, and through 6 months is assessed by Upper Leg Length (Thigh)/ Tibial Leg Length.
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 8 | 10 | 8
ratio
  Baseline: number analyzed (Participants) | 7 | 8 | 10 | 8
  Baseline | 1.089 (0.1067) | 1.074 (0.1350) | 1.107 (0.0607) | 1.061 (0.1341)
  Change from Baseline to Day 183: number analyzed (Participants) | 7 | 8 | 10 | 8
  Change from Baseline to Day 183 | 0.001 (0.0774) | 0.007 (0.0863) | 0.034 (0.1048) | 0.015 (0.1571)

19. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Tibial Length Ratio During Entire Study Period - Cohort 3 and 4
Description: The Upper Leg Length (Thigh) to Tibial Length Ratio prior to treatment, at baseline, and through 24 months is assessed by Upper Leg Length (Thigh)/ Tibial Leg Length.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 8
ratio
  Baseline | 1.107 (0.0607) | 1.061 (0.1341)
  Change from Baseline to Month 24 | 0.014 (0.0888) | -0.012 (0.1477)

20. Secondary Outcome: Change From Baseline in Upper Leg Length (Thigh) to Tibial Length Ratio During Entire Study Period - Cohort 1 and 2 Switchers
Description: as for outcome 19
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 6
ratio
  Baseline | 1.080 (0.1139) | 1.100 (0.1447)
  Change from Baseline to >=12 Months on 15ug/kg: number analyzed (Participants) | 3 | 6
  Change from Baseline to >=12 Months on 15ug/kg | -0.020 (0.0297) | 0.018 (0.1602)

21. Secondary Outcome: Change From Baseline in Arm Span to Height Ratio During Initial 6-months
Description: The Arm Span to Height Ratio prior to treatment, at baseline, and through 6 months is assessed by Arm Span / Standing Height.
Time Frame: At month 6 (Day 183)
Population: Efficacy Analysis Population
  Arm span measurement was optional until July 2015. Therefore data was not collected for all subjects for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 4 | 2 | 4 | 7
ratio
  Baseline | 0.901 (0.0189) | 0.889 (0.0906) | 0.913 (0.0123) | 0.893 (0.0284)
  Change from Baseline to Day 183 | 0.012 (0.0111) | -0.005 (0.0079) | 0.007 (0.0063) | 0.001 (0.0143)

22. Secondary Outcome: Change From Baseline in Arm Span to Height Ratio During Entire Study Period - Cohort 3 and 4
Description: The Arm Span to Height Ratio prior to treatment, at baseline, and through 24 months is assessed by Arm Span / Standing Height.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 8
ratio
  Baseline | 0.911 (0.0119) | 0.900 (0.0315)
  Change from Baseline to Month 24 | 0.000 (0.0123) | -0.006 (0.0290)

23. Secondary Outcome: Change From Baseline in Arm Span to Height Ratio During Entire Study Period - Cohort 1 and 2 Switchers
Description: The Arm Span to Height Ratio prior to treatment, at baseline, and through 24 months is assessed by Arm Span / Standing Height.
  Values are not available for participants in cohort 1 switchers for Change from Baseline to >=12 Months on 15ug/kg.
Time Frame: At month 24
Population: Efficacy Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 2
Number analyzed (Participants) | 6
ratio
  Baseline: number analyzed (Participants) | 5
  Baseline | 0.881 (0.0480)
  Change from Baseline to >=12 Months on 15ug/kg | -0.014 (0.0179)

ADVERSE EVENTS:
Time Frame: Up to Month 25 ± 7 Days
Description: Safety Analysis Population consists of all subjects who received at least one dose of study treatment and were used for safety analysis in the initial 6-month period and entire study period.
  Extension Safety Analysis Population consists of all subjects who received at least one dose of study treatment in the extension period and were used for safety analysis in the extension period.
Groups:
- Initial 6-Months Period 2.5 µg/kg.: BMN 111 at 2.5 μg/kg subcutaneous injection, once daily in the morning for initial 6-month period.
- Initial 6-Months Period 7.5 µg/kg.: BMN 111 at 7.5 μg/kg subcutaneous injection, once daily in the morning for initial 6-month period.
- Initial 6-Months Period 15 µg/kg.: BMN 111 at 15 μg/kg subcutaneous injection, once daily in the morning for initial 6-month period.
- Initial 6-Months Period 30 µg/kg.: BMN 111 at 30 μg/kg subcutaneous injection, once daily in the morning for initial 6-month period.
- Extension Period 2.5 µg/kg.: BMN 111 at 2.5 μg/kg subcutaneous injection, once daily in the morning for mean duration of 135.4 days.
- Extension Period 7.5 µg/kg.: BMN 111 at 7.5 μg/kg subcutaneous injection, once daily in the morning for mean duration of 83.1 days.
- Extension Period 15 µg/kg.: BMN 111 at 15 μg/kg subcutaneous injection, once daily in the morning for mean duration of 464.7 days.
- Extension Period 30 µg/kg.: BMN 111 at 30 μg/kg subcutaneous injection, once daily in the morning for mean duration of 546.4 days.
- Entire Study Period 2.5 µg/kg.: BMN 111 at 2.5 μg/kg subcutaneous injection, once daily in the morning for mean duration of 298.8 days.
- Entire Study Period 7.5 µg/kg.: BMN 111 at 7.5 μg/kg subcutaneous injection, once daily in the morning for mean duration of 175.5 days.
- Entire Study Period 15 µg/kg.: BMN 111 at 15 μg/kg subcutaneous injection, once daily in the morning for mean duration of 549.6 days.
- Entire Study Period 30 µg/kg.: BMN 111 at 30 μg/kg subcutaneous injection, once daily in the morning for mean duration of 650.9 days.
Arm/Group | Initial 6-Months Period 2.5 µg/kg. | Initial 6-Months Period 7.5 µg/kg. | Initial 6-Months Period 15 µg/kg. | Initial 6-Months Period 30 µg/kg. | Extension Period 2.5 µg/kg. | Extension Period 7.5 µg/kg. | Extension Period 15 µg/kg. | Extension Period 30 µg/kg. | Entire Study Period 2.5 µg/kg. | Entire Study Period 7.5 µg/kg. | Entire Study Period 15 µg/kg. | Entire Study Period 30 µg/kg.
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/9 | 0/7 | 0/14 | 0/22 | 0/8 | 0/8 | 0/15 | 0/22 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/9 | 1/7 | 0/14 | 1/22 | 1/8 | 1/8 | 0/15 | 1/22 | 1/9
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 10/10 | 9/9 | 7/7 | 13/14 | 22/22 | 8/8 | 8/8 | 14/15 | 22/22 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial 6-Months Period 2.5 µg/kg. (N=8) | Initial 6-Months Period 7.5 µg/kg. (N=8) | Initial 6-Months Period 15 µg/kg. (N=10) | Initial 6-Months Period 30 µg/kg. (N=9) | Extension Period 2.5 µg/kg. (N=7) | Extension Period 7.5 µg/kg. (N=14) | Extension Period 15 µg/kg. (N=22) | Extension Period 30 µg/kg. (N=8) | Entire Study Period 2.5 µg/kg. (N=8) | Entire Study Period 7.5 µg/kg. (N=15) | Entire Study Period 15 µg/kg. (N=22) | Entire Study Period 30 µg/kg. (N=9)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial 6-Months Period 2.5 µg/kg. (N=8) | Initial 6-Months Period 7.5 µg/kg. (N=8) | Initial 6-Months Period 15 µg/kg. (N=10) | Initial 6-Months Period 30 µg/kg. (N=9) | Extension Period 2.5 µg/kg. (N=7) | Extension Period 7.5 µg/kg. (N=14) | Extension Period 15 µg/kg. (N=22) | Extension Period 30 µg/kg. (N=8) | Entire Study Period 2.5 µg/kg. (N=8) | Entire Study Period 7.5 µg/kg. (N=15) | Entire Study Period 15 µg/kg. (N=22) | Entire Study Period 30 µg/kg. (N=9)
Injection site reaction (General disorders) | 2 | 6 | 8 | 9 | 2 | 5 | 15 | 6 | 2 | 8 | 17 | 9
Injection site erythema (General disorders) | 4 | 7 | 9 | 9 | 1 | 5 | 11 | 6 | 4 | 7 | 14 | 9
Injection site swelling (General disorders) | 4 | 2 | 4 | 2 | 0 | 0 | 8 | 1 | 4 | 2 | 8 | 2
Injection site urticaria (General disorders) | 1 | 1 | 2 | 3 | 1 | 1 | 3 | 1 | 1 | 2 | 3 | 4
Injection site pain (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 3
Pyrexia (General disorders) | 4 | 1 | 3 | 2 | 0 | 1 | 5 | 1 | 4 | 2 | 7 | 2
Injection site bruising (General disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0
Injection site pruritus (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3 | 1 | 0 | 1 | 4 | 2 | 1 | 3 | 7 | 2
Ear infection (Infections and infestations) | 0 | 3 | 2 | 2 | 1 | 1 | 4 | 2 | 1 | 4 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 5 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 2 | 1 | 0 | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 5 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 4 | 0 | 2 | 4 | 1 | 4 | 2 | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 3 | 3 | 2 | 2 | 4 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 1 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malpositioned teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 2 | 3 | 1 | 1 | 5 | 0 | 4 | 3 | 6 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 2 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Procedural anxiety (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 4 | 4 | 2 | 1 | 1 | 3 | 2 | 4 | 5 | 7 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 2 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 3 | 3 | 1
Ear swelling (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Blood immunoglobulin E increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep study abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Enuresis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Frustration tolerance decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Ear tube insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02055157/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT02055157/SAP_001.pdf